CLINICAL TRIAL: NCT00016315
Title: A Phase I Study of Gemcitabine, Carboplatin or Gemcitabine, Paclitaxel and Radiation Therapy Followed by Adjuvant Chemotherapy for Patients With Favorable Prognosis Inoperable Stage IIIA/B Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Gemcitabine, Carboplatin or Paclitaxel Plus Radiation Therapy in Treating Patients With Stage IIIA or IIIB Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0017; RTOG-L-0017; CDR0000068622
Record Dates: First submitted 2001-05-06; First posted 2003-05-07 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Gemcitabine; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (13):
- Arm 1 (Experimental): Sequence A: Gemcitabine 300 mg/m2/week plus radiation therapy (RT)
  Interventions: Drug: gemcitabine hydrochloride; Radiation: radiation therapy
- Arm 2 (Experimental): Sequence B: Gemcitabine 300 mg/m2/week plus paclitaxel 30 mg/m2/week and RT
  Interventions: Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: radiation therapy
- Arm 3 (Experimental): Sequence A: Gemcitabine 300 mg/m2/week plus carboplatin 2 AUC and RT
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride; Radiation: radiation therapy
- Arm 4 (Experimental): Sequence B: Gemcitabine 450 mg/m2/week plus paclitaxel 30 mg/m2/week and RT
  Interventions: Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: radiation therapy
- Arm 6 (Experimental): Sequence B: Gemcitabine 450 mg/m2/week plus paclitaxel 40 mg/m2/week and RT
  Interventions: Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: radiation therapy
- Arm 8 (Experimental): Sequence B: Gemcitabine 600 mg/m2/week plus paclitaxel 40 mg/m2/week and RT
  Interventions: Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: radiation therapy
- Arm 10 (Experimental): Sequence B: Gemcitabine 600 mg/m2/week plus paclitaxel 50 mg/m2/week and RT
  Interventions: Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: radiation therapy
- Arm 12 (Experimental): Sequence B: Gemcitabine 750 mg/m2/week plus paclitaxel 50 mg/m2/week and RT
  Interventions: Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: radiation therapy
- Arm 14 (Experimental): Sequence B: Gemcitabine 900 mg/m2/week plus paclitaxel 50 mg/m2/week and RT
  Interventions: Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: radiation therapy
- Arm 5 (Experimental): Sequence A: Gemcitabine 450 mg/m2/week plus carboplatin 2 AUC and RT
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride; Radiation: radiation therapy
- Arm 7 (Experimental): Sequence A: Gemcitabine 600 mg/m2/week plus carboplatin 2 AUC and RT
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride; Radiation: radiation therapy
- Arm 9 (Experimental): Sequence A: Gemcitabine 750 mg/m2/week plus carboplatin 2 AUC and RT
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride; Radiation: radiation therapy
- Arm 11 (Experimental): Sequence A: Gemcitabine 900 mg/m2/week plus carboplatin 2 AUC and RT
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin
  Arms: Arm 11; Arm 3; Arm 5; Arm 7; Arm 9
Drug: gemcitabine hydrochloride
Drug: paclitaxel
  Arms: Arm 10; Arm 12; Arm 14; Arm 2; Arm 4; Arm 6; Arm 8
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, carboplatin, and paclitaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining combination chemotherapy with radiation therapy in treating patients who have stage IIIA or stage IIIB non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of gemcitabine when administered with carboplatin and thoracic radiotherapy followed by adjuvant gemcitabine and carboplatin in patients with stage IIIA or IIIB non-small cell lung cancer.
* Determine the MTD of gemcitabine and paclitaxel when administered with thoracic radiotherapy followed by adjuvant gemcitabine and carboplatin in these patients.

OUTLINE: This is a multicenter, dose-escalation study of gemcitabine and paclitaxel. Patients are sequentially assigned to 1 of 3 treatment regimens.

* Regimen A: Patients receive gemcitabine IV over 30-60 minutes on days 1, 8, 22, 29, and 43 and thoracic radiotherapy daily 5 days a week for 7 weeks beginning on day 1.
* Regimen B (closed to accrual as of 5/13/03): Patients receive gemcitabine and thoracic radiotherapy as in regimen A and carboplatin IV over 30 minutes on days 1, 8, 22, 29, and 43.
* Regimen C: Patients receive gemcitabine and thoracic radiotherapy as in regimen A and paclitaxel IV over 1 hour on days 1, 8, 22, 29, and 43.

At 3 weeks after completion of chemoradiotherapy, all patients receive adjuvant gemcitabine IV over 30-60 minutes on days 71, 78, 92, and 99 and carboplatin IV over 30 minutes on days 71 and 92.

The first 6 patients enrolled receive regimen A to determine the safety of the initial dose of gemcitabine. After completion of regimen A, cohorts of 3-6 patients receive escalating doses of gemcitabine in regimen B (closed to accrual as of 5/13/03) until the maximum tolerated dose (MTD) is determined. In a separate sequence, cohorts of 3-6 patients receive alternating escalating doses of gemcitabine and paclitaxel in regimen C until the MTD is determined. The MTD is defined as the dose preceding that at which at least 3 of 6 patients experience dose-limiting toxicity.

Patients are followed at 3 months, 6 months, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 78 patients will be accrued for this study within 29 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed loco-regionally advanced non-small cell lung cancer meeting one of the following staging criteria:

  * Medically inoperable stage IIIA
  * Unresectable stage IIIA or IIIB
* Measurable disease on three-dimensional planning CT scan
* No post-resection intrathoracic tumor recurrence
* No pleural effusion on chest x-ray except those occurring after attempted thoracotomy or other invasive thoracic procedure
* No evidence of small cell histology
* No evidence of hematogenous or distant metastases

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least 100,000/mm^3
* Absolute granulocyte count at least 2,000/mm^3
* Hemoglobin at least 8.0 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* Serum glutamate oxaloacetate transaminase (SGOT) no greater than 1.5 times upper limit of normal (unless caused by documented benign disease)

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No myocardial infarction within the past 6 months
* No symptomatic heart disease, including angina, congestive heart failure, or uncontrolled arrhythmia

Pulmonary:

* Forced expiratory volume (FEV)_1 greater than 1,000 mL

Other:

* No other invasive malignancy within the past 3 years except nonmelanoma skin cancer
* No weight loss of more than 10% in 3 months prior to diagnosis
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior thoracic or neck radiotherapy

Surgery:

* See Disease Characteristics
* No prior complete or subtotal tumor resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2001-05; Primary Completion 2009-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of gemcitabine with carboplatin-based chemotherapy and radiation therapy | From start of treatment to 90 days
To determine the maximum tolerated dose of gemcitabine with paclitaxel-based chemotherapy and radiation therapy | From start of treatment to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Hak Choy, MD, Study Chair — Simmons Cancer Center
Locations (19):
- United States (19):
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - Monmouth Medical Center, Long Branch, New Jersey
  - Akron City Hospital, Akron, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Dale and Frances Hughes Cancer Center, East Stroudsburg, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin

REFERENCES:
- [Result] Choy H, Jain AK, Moughan J, Curran W, Whipple G, Demas WF, Ettinger DS. RTOG 0017: a phase I trial of concurrent gemcitabine/carboplatin or gemcitabine/paclitaxel and radiation therapy ("ping-pong trial") followed by adjuvant chemotherapy for patients with favorable prognosis inoperable stage IIIA/B non-small cell lung cancer. J Thorac Oncol. 2009 Jan;4(1):80-6. doi: 10.1097/JTO.0b013e318191503f. PMID 19096311
- [Result] Choy H, Swann S, Curran W, et al.: A phase I trial of gemcitabine, carboplatin or gemcitabine, paclitaxel and concurrent radiation therapy followed by consolidative gemcitabine and carboplatin for inoperable stage III non-small cell lung cancer: an RTOG 0017 study. [Abstract] Int J Radiat Oncol Biol Phys 63 (2 Suppl 1): A-70, S42, 2005.
- [Result] Choy H, Swann S, Walter C, et al.: A phase I trial of gemcitabine, carboplatin or gemcitabine, paclitaxel and concurrent radiation therapy followed by consolidative gemcitabine and carboplatin for inoperable stage III non-small cell lung cancer: an RTOG study. [Abstract] J Clin Oncol 23 (Suppl 16): A-7103, 646s, 2005.